CLINICAL TRIAL: NCT02455089
Title: Prognosis Assessment of the Increase of GADD34 Gene Expression for Patient Suffering From Systemic Lupus Erythematosus
Acronym: GADD34-LES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 38RC15.010; 2015-A00493-46 (Other: ID RCB)
Record Dates: First submitted 2015-04-21; First posted 2015-05-27 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Lupus Erythematosus
Keywords: Flare; Therapeutic adjustments; Biological Marker; Immunologic Marker; Prognosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Test group (Experimental): 250 SLE patients : All SLE patients included in the study. Intervention : Blood analysis including GADD34 RNA level measurement every 3 months up to 1 year.
  They will provided a blood sample every 3 months during a year. The result of GADD34 RNA level in mononuclear blood cells will be correlated to the clinical assessment of a SLE flare during the next 3 months.
  A flare occurence will the group
  Interventions: Other: GADD34 RNA level measurement.

INTERVENTIONS:
Other: GADD34 RNA level measurement. — Blood analysis including GADD34 RNA level measurement is performed every 3 months up to 1 year for SLE patients.
  A modal including physical exam, standard biological results and GADD34 RNA level is correlated to a SLE flare occurence in the next 3 months.
  Other Names: Experimental: Test group

SUMMARY:
Given that GADD34 has been described as a potential key regulator of pro-inflammatory cytokine production in human and elevated blood marker in SLE patients, this study aim to prove that the GADD34 RNA level in mononuclear blood cells can be used as a prognostic marker to assess the risk of SLE flare.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) has a prevalence estimated between 1 and 6 per 10000 individuals and concerns over 30 000 patients in France for example. As of today, there isn't any reliable specific blood analysis that can be used to assess the prognosis of SLE, that means predict a SLE flare. The discovery of such a blood test could allow a better patients' monitoring in order to help doctors to better adapt treatments (lowering background treatments when they are not needed and increase them ahead of a potential flare when the risk assessment raises).

In SLE patients, a recent study shows elevated levels of GADD34 RNA in mononuclear blood cells : higher than twice the control levels for 36 of the 60 SLE patients and ten times higher than the control levels for 13 of the 60 SLE patients.

Given that GADD34 has been described as a potential key regulator of pro-inflammatory cytokine production in human and elevated blood marker in SLE patients, this study aim to prove that the GADD34 RNA level in mononuclear blood cells can be used as a prognostic marker to assess the risk of SLE flare.

ELIGIBILITY:
* Inclusion Criteria:

  * man and women over 18 Years old.
  * suffering from SLE (American College of Rheumatology criteria).
  * without SLE flare for 3 months.
  * with a signed consent and social security affiliation (required in France).
* Exclusion Criteria:

  * Viral infection within 15 days.
  * Other chronic inflammatory disease.
  * People with special protection (defined in articles : L1121- §5-8 et articles L3212-§1-3 of French health care law).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
GADD34 RNA level | Measured every 3 months, up to 1 year (5 blood samples).The Last result before a SLE flare occurence will be used.
  GADD34 RNA level in mononuclear blood cells in the last 3 months before a SLE flare occurence.
  RNA levels have no unit,they are rates compared with a housekeeping gene RNA level as unit.
  To avoid any bias in primary outcome, SLE Flare occurence is assessed with both patient and investigator blinded from Gadd34 RNA level.

SECONDARY OUTCOMES:
Prognosis score of SLE flare occurence | Measured every 3 months, up to 1 year (5 blood samples).The Last result before a SLE flare occurence will be used.
  Prognosis score of SLE flare occurence using a modal including GADD34 RNA increase, SLEDAI score and Physician Global Assessment (PGA).
  This modal is compared to the gold standard modal which use only PGA and SLEDAI Score in term of sensibility and specificity.
Pro-inflammatory cytokine blood level. | Measured every 3 months, up to 1 year (5 blood samples).
  Correlation between GADD34 RNA increase or decrease and interferon-alpha, interferon-beta, interleukin-6 and interleukine-17 levels.

OTHER OUTCOMES:
GADD34 RNA level in each mononuclear blood cells (B cells, T cells and monocytes). | Measured once at the 2nd visit (3 months after the inclusion).
  GADD34 RNA level is measured respectively in B cells, T cells and monocytes and is compared with each other.
  RNA levels have no unit,they are rates compared with a housekeeping gene RNA level as unit. This outcome is measured only for 30 patients.
GADD34 RNA level in non-mononuclear blood cells | Measured once at the 2nd visit (3 months after the inclusion).
  GADD34 RNA level is measured respectively in non-mononuclear blood cells and is compared with GADD34 RNA level in mononuclear blood cells.
  RNA levels have no unit,they are rates compared with a housekeeping gene RNA level as unit. This outcome is measured only for 30 patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves Cesbron, MD, Principal Investigator — University Hospital of Grenoble, France.
Locations (7):
- France (7):
  - CHU Grenoble, Grenoble
  - groupement hospitalier mutualiste de Grenoble, Grenoble
  - Hopital européen de Marseille, Marseille
  - CHU Marseille, Marseille
  - CHR Annecy Genevois, Metz-Tessy
  - CHU Lyon sud, Pierre-Bénite
  - CHU Saint Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: Yes
No data will be be shared with non associated investigator till publication. Possibility to share after publication, through formol requirement adressed to Grenoble hospital administration (AccueilRecherche@chu-grenoble.fr)

REFERENCES:
- [Result] Claudio N, Dalet A, Gatti E, Pierre P. Mapping the crossroads of immune activation and cellular stress response pathways. EMBO J. 2013 May 2;32(9):1214-24. doi: 10.1038/emboj.2013.80. Epub 2013 Apr 12. PMID 23584529
- [Result] Clavarino G, Claudio N, Couderc T, Dalet A, Judith D, Camosseto V, Schmidt EK, Wenger T, Lecuit M, Gatti E, Pierre P. Induction of GADD34 is necessary for dsRNA-dependent interferon-beta production and participates in the control of Chikungunya virus infection. PLoS Pathog. 2012;8(5):e1002708. doi: 10.1371/journal.ppat.1002708. Epub 2012 May 17. PMID 22615568
- [Result] Clavarino G, Claudio N, Dalet A, Terawaki S, Couderc T, Chasson L, Ceppi M, Schmidt EK, Wenger T, Lecuit M, Gatti E, Pierre P. Protein phosphatase 1 subunit Ppp1r15a/GADD34 regulates cytokine production in polyinosinic:polycytidylic acid-stimulated dendritic cells. Proc Natl Acad Sci U S A. 2012 Feb 21;109(8):3006-11. doi: 10.1073/pnas.1104491109. Epub 2012 Feb 6. PMID 22315398
- [Result] Costedoat-Chalumeau N, Galicier L, Aumaitre O, Frances C, Le Guern V, Liote F, Smail A, Limal N, Perard L, Desmurs-Clavel H, Boutin du LT, Asli B, Kahn JE, Pourrat J, Sailler L, Ackermann F, Papo T, Sacre K, Fain O, Stirnemann J, Cacoub P, Jallouli M, Leroux G, Cohen-Bittan J, Tanguy ML, Hulot JS, Lechat P, Musset L, Amoura Z, Piette JC; Group PLUS. Hydroxychloroquine in systemic lupus erythematosus: results of a French multicentre controlled trial (PLUS Study). Ann Rheum Dis. 2013 Nov;72(11):1786-92. doi: 10.1136/annrheumdis-2012-202322. Epub 2012 Nov 10. PMID 23144449
- [Result] Niewold TB, Clark DN, Salloum R, Poole BD. Interferon alpha in systemic lupus erythematosus. J Biomed Biotechnol. 2010;2010:948364. doi: 10.1155/2010/948364. Epub 2010 Jun 29. PMID 20652065
- [Result] Novoa I, Zeng H, Harding HP, Ron D. Feedback inhibition of the unfolded protein response by GADD34-mediated dephosphorylation of eIF2alpha. J Cell Biol. 2001 May 28;153(5):1011-22. doi: 10.1083/jcb.153.5.1011. PMID 11381086
- [Result] Petri MA, van Vollenhoven RF, Buyon J, Levy RA, Navarra SV, Cervera R, Zhong ZJ, Freimuth WW; BLISS-52 and BLISS-76 Study Groups. Baseline predictors of systemic lupus erythematosus flares: data from the combined placebo groups in the phase III belimumab trials. Arthritis Rheum. 2013 Aug;65(8):2143-53. doi: 10.1002/art.37995. PMID 23754628
- [Result] Ronnelid J, Tejde A, Mathsson L, Nilsson-Ekdahl K, Nilsson B. Immune complexes from SLE sera induce IL10 production from normal peripheral blood mononuclear cells by an FcgammaRII dependent mechanism: implications for a possible vicious cycle maintaining B cell hyperactivity in SLE. Ann Rheum Dis. 2003 Jan;62(1):37-42. doi: 10.1136/ard.62.1.37. PMID 12480667
- [Result] Wang S, Kaufman RJ. The impact of the unfolded protein response on human disease. J Cell Biol. 2012 Jun 25;197(7):857-67. doi: 10.1083/jcb.201110131. PMID 22733998
- [Result] Yap DY, Lai KN. The role of cytokines in the pathogenesis of systemic lupus erythematosus - from bench to bedside. Nephrology (Carlton). 2013 Apr;18(4):243-55. doi: 10.1111/nep.12047. PMID 23452295